CLINICAL TRIAL: NCT01966978
Title: The Effect of Simple Insulin Detemir Titration, Metformin Plus Liraglutide Compared to Simple Insulin Detemir Titration Plus Insulin Aspart and Metformin for Type 2 Diabetes With Very Elevated HbA1c - The SIMPLE Study: A 26 Week, Randomized, Open Label, Parallel-group, Intention to Treat Study
Brief Title: The Effect of Simple Basal Insulin Titration, Metformin Plus Liraglutide for Type 2 Diabetes With Very Elevated HbA1c - The SIMPLE Study
Acronym: SIMPLE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Ildiko Lingvay, MD, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STU 072013-030
Record Dates: First submitted 2013-10-17; First posted 2013-10-22 (Estimated); Results first posted 2019-10-22 (Actual); Last update posted 2019-10-22 (Actual); Status verified 2019-10

CONDITIONS: Diabetes Mellitus, Type 2; Diabetes
Keywords: Diabetes Mellitus, Type 2; Insulin; Insulin, Long-Acting; Insulin, Short Acting; Detemir; Liraglutide; GLP-1; Glucagon Like Peptide; Metformin; Uncontrolled Diabetes; Elevated A1c; Incretins
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus; Insulin Resistance | interventions — Metformin; Insulin Detemir; Liraglutide; Insulin Aspart

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control: Metformin, Insulin Detemir, Insulin Aspart (Active Comparator): Metformin titrated to max tolerated dose (at least 1000 mg/day); Insulin detemir titrated based on the study protocol; Insulin Aspart titrated by the physician
  Interventions: Drug: Metformin; Drug: Detemir; Drug: Insulin Aspart
- Metformin, insulin determir, Liraglutide (Active Comparator): Metformin titrated to max tolerated dose (at least 1000mg/day); Insulin detemir titrated based on the study protocol"; Liraglutide titrated to max tolerated dose (at least 1.2 mg/day)
  Interventions: Drug: Metformin; Drug: Detemir; Drug: Liraglutide

INTERVENTIONS:
Drug: Metformin — Metformin will be started at 500 mg daily (or continued at current dose)and weekly titrated to 2000 mg or maximum tolerated dose (at least 1000 mg/day)
  Other Names: Metformin tablets
Drug: Detemir — Insulin detemir will be started in both groups at 0.3 units/kg or conversion 1:1 from dose of basal insulin prior to randomization. The titration will be primarily patient-driven, based on our study protocol table. Additional physician driven titration will be allowed in both groups if patient fails to intensify basal insulin dose as directed.
  Other Names: Insulin Detemir subcutaneous once or twice daily
Drug: Liraglutide — Initial dose of 0.6 mg/day with weekly increments of 0.6 mg until dose of 1.8 mg/day or maximal tolerated dose (at least 1.2 mg/day)is reached
  Other Names: Liraglutide 6 mg/mL Subcutaneously
  Arms: Metformin, insulin determir, Liraglutide
Drug: Insulin Aspart — Insulin aspart will be initiated at a dose of 0.3 units/kg/day divided among the number of meals taken daily and titrated based on physician clinical judgment with the goal of pre-prandial BG 70-130 mg/dL and post-prandial BG <180
  Other Names: Insulin Aspart Subcutaneous injection one to three times daily
  Arms: Control: Metformin, Insulin Detemir, Insulin Aspart

SUMMARY:
The aim of this clinical trial is to assess and compare the effect of insulin detemir in combination with liraglutide and metformin versus insulin detemir in combination with insulin aspart and metformin in subjects with very uncontrolled Type 2 Diabetes (A1c > 10%).

DETAILED DESCRIPTION:
The aim of this study is to compare a GLP-1 plus basal insulin and metformin treatment regimen to a basal-bolus plus metformin treatment regimen in patients with very uncontrolled (HbA1c>10%) type 2 diabetes. The investigators will compare the two regimens with respect to efficacy in improving glycemic control, rate of hypoglycemia, change in weight, effect on patient quality of life, treatment burden, physician time, as well as healthcare related cost. The investigators hypothesize that at 26 weeks from randomization the two treatment regimens will have similar percentage of patients reaching A1c levels <7.0%, while more patients on the GLP-1 plus basal insulin strategy will achieve the composite end point of A1c levels <7.0% without severe hypoglycemia or significant weight gain.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis of type 2 diabetes with confirmed HbA1c level >10% at time of enrollment, regardless of prior or current treatment regimens, or time since diagnosis.

Exclusion Criteria:

1. Age <18 as the feasibility and safety of this treatment regimen should be first established in the adult population; if successful, a subsequent pediatric study will be proposed;
2. Type 1 diabetes as purposefully withholding meal-time insulin is contraindicated;
3. Clinical state requiring inpatient admission/treatment;
4. Contraindication or strong cautions to any of the study medications:

   1. Creatinine above 1.4 mg/dl for women and 1.5 mg/dl for men (per metformin label)
   2. History of lactic acidosis (per metformin label)
   3. Advanced hepatic or cardiac disease (per metformin label)
   4. Age >80 years (per metformin label)
   5. Chronic alcohol use (>14 drinks/week)
   6. History of pancreatitis (per liraglutide label)
   7. Personal or family history of medullary thyroid cancer or MEN syndrome (per liraglutide label)
   8. Pregnancy and lactation (per liraglutide label)
5. Any serious or unstable medical condition as it would interfere with treatment assignment as well as outcome measurement;
6. Any scheduled elective procedures/surgeries;
7. Active infections, including osteomyelitis;
8. Not willing to participate, unable to keep projected appointments, unwillingness to receive injectable treatment; unwillingness to perform 7-point glucose profiles over 2 consecutive days the weeks prior to Randomization (visit 1)and the week prior to visit 6
9. Non English speaking.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 157 (Actual)
Dates: Start 2014-11; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ildiko Lingvay, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- UT Southwestern Medical Center, Dallas, Texas, United States

REFERENCES:
- [Derived] Patel S, Abreu M, Tumyan A, Adams-Huet B, Li X, Lingvay I. Effect of medication adherence on clinical outcomes in type 2 diabetes: analysis of the SIMPLE study. BMJ Open Diabetes Res Care. 2019 Nov 18;7(1):e000761. doi: 10.1136/bmjdrc-2019-000761. eCollection 2019. PMID 31803482

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Total number of subjects consented is 157, total number of subjects randomized is 120, of those 120 only 110 are MITT data set
Period: Overall Study
Arm/Group | Control: Metformin, Insulin Detemir, Insulin Aspart | Metformin, Insulin Determir, Liraglutide
Started | 61 | 59
Completed | 44 | 46
Not Completed | 17 | 13

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control: Metformin, Insulin Detemir, Insulin Aspart | Metformin, Insulin Determir, Liraglutide | Total
Number analyzed (Participants) | 61 | 59 | 120
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.1 (10.0) | 46.7 (9.0) | 47.4 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45 | 40 | 85
  Male | 16 | 19 | 35
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic | 21 | 27 | 48
  Non-Hispanic White | 10 | 12 | 22
  African-American | 30 | 20 | 50
HbA1c [Mean (Standard Deviation); unit: percentage of glycosylated hemoglobin] | 12.0 (1.5) | 12.1 (1.4) | 12.1 (1.4)

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Randomization in A1c at Week 26
Description: Change in glycosylated Hemoglobin A1c (A1c) from randomization to 26 weeks of therapy
Time Frame: Baseline and Week 26
Measure: Mean (95% Confidence Interval); unit: Percentage of glycosylated hemoglobin
Arm/Group | Control: Metformin, Insulin Detemir, Insulin Aspart | Metformin, Insulin Determir, Liraglutide
Number analyzed (Participants) | 44 | 46
Percentage of glycosylated hemoglobin | 3.4 [2.4 to 3.7] | 4.1 [3.5 to 4.8]

2. Secondary Outcome: Composite End-point
Description: Percentage of participants with glycosylated Hemoglobin A1c (A1c)<8% AND no documented severe hypoglycemia (<56 mg/dL) during the study AND no significant weight gain (>3% from baseline)
Time Frame: Week 0 (Randomization) , Week 26
Measure: Number; unit: percentage of participants
Arm/Group | Control: Metformin, Insulin Detemir, Insulin Aspart | Metformin, Insulin Determir, Liraglutide
Number analyzed (Participants) | 44 | 46
percentage of participants | 16 | 34

3. Secondary Outcome: Percentage of Participants Reaching Target A1c of <7% at Week 26
Time Frame: Week 26
Measure: Number; unit: percentage of participants
Arm/Group | Control: Metformin, Insulin Detemir, Insulin Aspart | Metformin, Insulin Determir, Liraglutide
Number analyzed (Participants) | 44 | 46
percentage of participants | 20 | 44

4. Secondary Outcome: Percentage of Participants Reaching Pre-specified "Treatment Failure" Outcome
Description: Treatment Failure defined as A1c>10% at week 13 (visit 5)
Time Frame: week 13
Measure: Number; unit: percentage of participants
Arm/Group | Control: Metformin, Insulin Detemir, Insulin Aspart | Metformin, Insulin Determir, Liraglutide
Number analyzed (Participants) | 44 | 46
percentage of participants | 16.1 | 7.4

5. Secondary Outcome: Mean Change From Randomization in Body Weight
Description: Change in body weight from randomization to end of study.
Time Frame: Week 0 (Randomization) , Week 26
Measure: Mean (95% Confidence Interval); unit: kilogram
Arm/Group | Control: Metformin, Insulin Detemir, Insulin Aspart | Metformin, Insulin Determir, Liraglutide
Number analyzed (Participants) | 44 | 46
kilogram | 3.1 [1.7 to 4.6] | -0.6 [-0.9 to 2.1]

6. Secondary Outcome: Hypoglycemic Episodes
Description: Percentage of participants experiencing any episodes of documented hypoglycemia defined as CBG reading of <70 mg/dl
Time Frame: Week 0 (Randomization) , Week 2, week 4, week 13, Week 26
Measure: Number; unit: percentage of participants
Arm/Group | Control: Metformin, Insulin Detemir, Insulin Aspart | Metformin, Insulin Determir, Liraglutide
Number analyzed (Participants) | 44 | 46
percentage of participants | 66.1 | 35.2

7. Secondary Outcome: Change in Diabetes Quality of Life (DQOL)Questionnaire Score- Least Squares Means
Description: Diabetes Quality of Life (DQOL) questionnaires will be completed by the patient at the randomization and end-of study visits. ALL D-QOL domains are scored on a 1-5 scale, with a lower number representing better quality of life or treatment satisfaction. Outcome reported is difference between mean baseline and mean Week 26 score.
Time Frame: Week 0 (Randomization) , Week 26
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Control: Metformin, Insulin Detemir, Insulin Aspart | Metformin, Insulin Determir, Liraglutide
Number analyzed (Participants) | 44 | 46
score on a scale
  General Health Perception | -0.3 [-0.6 to -0.1] | -0.9 [-1.1 to -0.6]
  Current Health Perception | -0.5 [-0.9 to -0.1] | -1.1 [-1.5 to -0.7]
  Treatment Satisfaction | -0.3 [-0.5 to -0.04] | -0.6 [-0.8 to -0.4]
  Diabetes Related Worry | 0.03 [-0.1 to 0.2] | -0.2 [-0.4 to -0.04]
  Social or Vocational Worry | -0.02 [-0.3 to 0.3] | -0.2 [-0.4 to 0.08]
  Hypoglycemia Fear | 0.3 [0.04 to 0.5] | -0.2 [-0.4 to -0.005]
  Glycemic Control Perception | -1.1 [-1.6 to -0.7] | -1.6 [-2.0 to -1.2]
  Satisfaction with Insulin Treatment | -1.3 [-1.8 to -0.8] | -1.7 [-2.2 to -1.2]
  Willingness to Continue Insulin Treatment | -0.9 [-1.4 to -0.3] | -1.1 [-1.7 to -0.6]
  LifeStyle Flexibility | -0.09 [-0.4 to 0.2] | -0.2 [-0.4 to 0.1]
  Social Stigma | 0.1 [-0.2 to 0.4] | 0.01 [-0.3 to 0.4]

8. Secondary Outcome: Change in Short Form-36 (SF-36) Questionnaire Score
Description: Quality of life questionnaires will be completed by the patient at the randomization and end-of study visits. SF-36 is scored on a 1-100 scale; a higher score represents a better self-assessed health - for all domains.
Time Frame: Week 0 (Randomization) , Week 26
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Control: Metformin, Insulin Detemir, Insulin Aspart | Metformin, Insulin Determir, Liraglutide
Number analyzed (Participants) | 44 | 46
score on a scale
  Physical Component Summary | -0.1 [-0.4 to 0.2] | 0.007 [-0.3 to 0.3]
  Mental Component Summary | 0.04 [-0.1 to 0.1] | 0.09 [-0.02 to 0.2]

ADVERSE EVENTS:
Time Frame: 6 months (Baseline to Week 26)
Description: Adverse events were collected both by self-report as well as review of the electronic health record. Nausea, vomiting, headache, diarrhea and abdominal pain were pre-defined events of special interest and proactively elicited at each visit from all patients.
Arm/Group | Control: Metformin, Insulin Detemir, Insulin Aspart | Metformin, Insulin Determir, Liraglutide
All-Cause Mortality (participants affected / at risk) | 0/56 | 0/54
Serious Adverse Events (participants affected / at risk) | 13/56 | 6/54
Other Adverse Events (participants affected / at risk) | 40/56 | 50/54
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Control: Metformin, Insulin Detemir, Insulin Aspart (N=56) | Metformin, Insulin Determir, Liraglutide (N=54)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Facial Burn (Skin and subcutaneous tissue disorders) | 1 | 0
Urinary Tract Infection (Renal and urinary disorders) | 1 | 0
Respiratory Distress (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 | 1
Small Bowel Obstruction (Gastrointestinal disorders) | 1 | 0
Fall (Investigations) | 2 | 0
chest pain (Cardiac disorders) | 0 | 1
Diabetic Ketoacidosis (Endocrine disorders) | 4 | 0
Osteomyelitis (Musculoskeletal and connective tissue disorders) | 1 | 0
hypertension (Cardiac disorders) | 0 | 1
myocardial infarction (Cardiac disorders) | 1 | 1
nasopharyngeal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
psychiatric inpatient hospitalization (Psychiatric disorders) | 0 | 1
vitreal hemmorhage (Eye disorders) | 0 | 1
bacteremia (Infections and infestations) | 1 | 0
puncture wound (Injury, poisoning and procedural complications) | 1 | 0
nephrotic syndrome (Renal and urinary disorders) | 1 | 0
Lower GI bleed (Gastrointestinal disorders) | 1 | 0
glaucoma (Eye disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Control: Metformin, Insulin Detemir, Insulin Aspart (N=56) | Metformin, Insulin Determir, Liraglutide (N=54)
headache (Nervous system disorders) | 10 | 14
GI (Gastrointestinal disorders) | 28 | 42
Other AE (Investigations) | 9 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-05-06): https://cdn.clinicaltrials.gov/large-docs/78/NCT01966978/Prot_SAP_000.pdf